CLINICAL TRIAL: NCT01784029
Title: Comparison of Two Standard High-dose Treatment Regimens for Vitamin D Deficiency in Minority Adolescents: Associations of Vitamin D Repletion With Changes in Markers of Musculoskeletal, Cardiometabolic, and Immune Function
Brief Title: Treatment Study of Vitamin D Deficiency in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Susan Coupey, Chief, Adolescent Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-09-345
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Vitamin D Deficiency
Keywords: adolescents; minority
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Experimental): VItamin D3 1,000 IU
  1 x day, 8 weeks
  Interventions: Drug: Vitamin D3
- Weekly High Dose (Experimental): Vitamin D3 50,000 IU
  1x week, 8 weeks
  Interventions: Drug: Vitamin D3
- Daily High Dose (Experimental): Vitamin D3 5,000 IU
  1x day, 8 weeks
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Doses are as mentioned above. Will repeat 3 month cycles of treatment if still deficient at 3 month follow up.
  Other Names: cholecalciferol

SUMMARY:
To compare the efficacy of two high dose vitamin D3 regimens (5,000 IU daily vs. 50,000 IU weekly) used clinically for the treatment of vitamin D deficiency versus a low dose of vitamin D3 used for supplementation (1,000 IU daily) in a clinical sample of predominantly Hispanic and black adolescents with vitamin D deficiency [25(OH)D level <20 ng/ml] by assessing change in 25(OH)D levels before and after 8 weeks of treatment.

To compare the effects of vitamin D repletion [25(OH)D level >20 ng/mL] on selected musculoskeletal, cardiometabolic and immune markers in predominantly Hispanic and black adolescents with vitamin D deficiency [25(OH)D level < 20 ng/mL].

Hypothesis 1: Increase in vitamin D level will be associated with improvement in musculoskeletal, cardiometabolic, and immune markers including blood pressure, waist circumference, musculoskeletal symptoms, asthma severity and hand-grip strength.

DETAILED DESCRIPTION:
Vitamin D is an essential nutrient and pro-hormone that has garnered widespread attention over the past decade for both its known and theorized health benefits. Patients, clinicians and researchers have all been alerted to the increasing prevalence of vitamin D deficiency (defined as level of 25(OH)D <20 ng/mL) and the significance of the extra-skeletal health effects of vitamin D. Aside from the skeletal impacts of Vitamin D, there has been recent evidence about potential health benefits of vitamin D related to the multiple extra-skeletal roles of this hormone. In fact, vitamin D receptors are found in many organs including brain, heart, skin, small intestine, gonads, prostate and breast as well in almost all nucleated cells including osteoblasts, activated T and B-lymphocytes, and B islet cells. Studies in children and adolescents as well as in adults show associations of vitamin D deficiency with cardiovascular risk factors, musculoskeletal health, asthma, and autoimmune diseases.

While Vitamin D deficiency is quite prevalent, adolescents who are obese or who are darker skinned are consistently shown to have higher rates of vitamin D deficiency than lean and lighter skinned adolescents. Treatment of vitamin D deficiency and maintenance of sufficient levels in adolescents are largely under-studied leaving patients and clinicians without clear evidence-based guidelines to follow.

The goal of this study is to compare the efficacy of different treatment regimens for vitamin D deficiency in our population of predominantly minority adolescents and to examine the effect of correction of vitamin D deficiency on selected extra-skeletal targets of vitamin D action including musculoskeletal, cardiometabolic, and immune function.

ELIGIBILITY:
Inclusion Criteria:

* age 13-20

Exclusion Criteria:

* currently receiving treatment for hypovitaminosis D
* hepatic or renal disease
* metabolic rickets
* inability to complete the questionnaire

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Coupey, MD, Principal Investigator — Children's Hospital at Montefiore
Locations (1):
- Children's Hospital at Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Talib HJ, Ponnapakkam T, Gensure R, Cohen HW, Coupey SM. Treatment of Vitamin D Deficiency in Predominantly Hispanic and Black Adolescents: A Randomized Clinical Trial. J Pediatr. 2016 Mar;170:266-72.e1. doi: 10.1016/j.jpeds.2015.11.025. Epub 2015 Dec 18. PMID 26707619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited aged 13-20 years from the Adolescent Medicine and Pediatric Endocrinology practices at Children's Hospital at Montefiore.
Pre-assignment Details: Of the 305 adolescents screened, only 203 met the inclusion criteria of being vitamin D deficient. Of the 203 adolescents identified with vitamin D deficiency, 20 were unable to be further contacted and randomized.
Groups:
- Low Dose: VItamin D3 1,000 IU
  1 x day, 8 weeks
  Vitamin D3: Doses are as mentioned above. Will repeat 3 month cycles of treatment if still deficient at 3 month follow up.
- Weekly High Dose: Vitamin D3 50,000 IU
  1x week, 8 weeks
  Vitamin D3: Doses are as mentioned above. Will repeat 3 month cycles of treatment if still deficient at 3 month follow up.
- Daily High Dose: Vitamin D3 5,000 IU
  1x day, 8 weeks
  Vitamin D3: Doses are as mentioned above. Will repeat 3 month cycles of treatment if still deficient at 3 month follow up.
Period: Overall Study
Arm/Group | Low Dose | Weekly High Dose | Daily High Dose
Started | 61 | 59 | 63
Completed | 42 | 39 | 41
Not Completed | 19 | 20 | 22
Not completed — Lost to Follow-up | 19 | 20 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | Weekly High Dose | Daily High Dose | Total
Number analyzed (Participants) | 61 | 59 | 63 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (2.1) | 16.5 (2.4) | 16.6 (2.1) | 16.6 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 46 | 136
  Male | 16 | 14 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in 25(OH)D Serum Level After Treatment for Vitamin D Deficiency (Deficiency Defined as 25(OH)D <20 ng/dL)
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low Dose | Weekly High Dose | Daily High Dose
Number analyzed (Participants) | 42 | 39 | 41
ng/mL | 6.2 (6.5) | 24.9 (15.1) | 21 (15.2)

ADVERSE EVENTS:
Time Frame: Duration of study (1 year)
Arm/Group | Low Dose | Weekly High Dose | Daily High Dose
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59 | 0/63
Other Adverse Events (participants affected / at risk) | 0/61 | 0/59 | 0/63

LIMITATIONS AND CAVEATS:
Substantial attrition rate is a limitation of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No